RAPID local ischemic postconditioning in acute ischemic Stroke
pAtients receiVEd successful thrombectomy reperfusion (RAPID-SAVE)

# STATISTICAL ANALYSIS PLAN

# Principal Investigator

Yueqi Zhu, MD, PhD

Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

Clinical Trial: NCT06526429

Protocol Version 1.0

Oct 14, 2024

| 1 | <b>BOIN12 Study Design and Statistical Analysis Plan</b> |
|---|---|
| 2 | This study employed the Bayesian optimal interval phase I/II (BOIN12) trial design <sup>1</sup> |
| 3 | find the optimal biological dose (OBD). The BOIN12 design used utility to quantify |
| 4 | the desirability of a dose in terms of toxicity-efficacy trade off and adaptively |
| 5 | allocated patients to the dose that has the highest estimated desirability. The utilities |
| 6 | ascribed to each possible efficacy-toxicity outcome were as follows: (No Toxicity, |
| 7 | Efficacy) = 100; (Toxicity, Efficacy) = 60; (No Toxicity, No Efficacy) = 40; and |
| 8 | (Toxicity, No Efficacy) = 0. A higher value indicated a more desirable outcome (0 |
| 9 | and 100 present the least and most desirable outcome, respectively). |
| 10 | Let $u1,\dots,u4$ denoted these utilities. Given a dose $j$ , let $p1,\dots,p4$ denoted the |
| 11 | corresponding probabilities of observing each of the possible toxicity-efficacy |
| 12 | outcomes. Then, the mean utility of dose $j$ is |
| 13 | uj=p1u1+p2u2+p3u3+p4u4. |
| 14 | A higher value of $uj$ indicated a higher desirability of dose $j$ in terms of risk-benefit |
| 15 | tradeoff. To safeguard patients from toxic and/or futile doses, two dose acceptability |
| 16 | criteria were used by BOIN12 to decide which doses might be used to treat patients. |
| 17 | A dose was deemed as admissible and eligible for treating patients if it satisfied the |
| 18 | following safety and efficacy criteria. |
| 19 | (Safety) Pr( $(\pi T > 0.15 data)$ ) < 0.95, |
| 20 | (Efficacy) $Pr(\pi E < 0.6 data) < 0.9$ . |
| 21 | where $\pi T$ and $\pi E$ were the true DLT rate and efficacy rate, respectively. These two |
| 22 | conditions ensured that the admissible dose could not be overly toxic or futile. Doses |
| 23 | that were not admissible would be eliminated from the trial. If a dose was eliminated |
| 24 | due to toxicity, all doses higher than that dose would also be eliminated. The |
| 25 | objective was to identify the OBD, defined as the dose that was admissible and had |
| 26 | the highest desirability. |

| 27 | We planned to enrol a maximum number of 60 patients with a cohort size of 5. When |
|---|---|
| 28 | the current dose's observed toxicity rate fell within the stay interval of BOIN, we |
| 29 | would stop exploring higher doses if its number of patients $\ge N*$ , where $N*=5$ . The |
| 30 | BOIN12 design is depicted in Supplemental Figure 1 and it was implemented |
| 31 | according to the following 3 steps via the BOIN12 shiny app <sup>2</sup> . |
| 32 | 1. Treat the first cohort at dose level 3. |
| 33 | 2. Suppose that the current dose level is $j$ , choose one of the following three |
| 34 | cases to determine the dose for treating the next cohort of patients: |
| 35 | Case A: determine the desirability of dose levels $j-1$ , $j$ , and $j+1$ using the |
| 36 | rank-based desirability score (RDS) table (Table 1), and choose the one that |
| 37 | has the highest desirability to treat the next cohort. If the RDS of all three |
| 38 | doses are "E," stop the trial and no dose should be selected. In the case that |
| 39 | dose level $j-1$ (or $j+1$ ) does not exist, then apply the above rule to dose |
| 40 | levels $j$ and $j+1$ (or $j$ and $j-1$ ). |
| 41 | Case B: determine the desirability of dose levels $j$ and $j-1$ using the RDS |
| 42 | table (Table 1), and choose the one that has the higher desirability to treat the |
| 43 | next cohort. If the RDS of the two doses are "E," stop the trial and no dose |
| 44 | should be selected. If the current dose level $j$ is the lowest dose, treat the next |
| 45 | cohort of patients at the lowest dose unless the RDS of the lowest dose is "E," |
| 46 | at which point terminate the trial. |
| 47 | Case C: determine the desirability of dose levels $j$ and $j-1$ using the RDS |
| 48 | table (Table 1). |
| 49 | $\circ$ If the current dose level $j$ is the lowest dose, treat the new patients at |
| 50 | the lowest dose unless the RDS of the lowest dose is "E," at which |
| 51 | point terminate the trial. |

| 52 | $\circ$ If the current dose level $j$ is not the lowest dose and the RDS of dose |
|---|---|
| 53 | level $j-1$ is not "E," de-escalate the dose to level $j-1$ to treat the next |
| 54 | cohort of patients. |
| 55 | If the current dose level $j$ is not the lowest dose and the RDS of dose |
| 56 | level $j-1$ is "E," stay at the current dose level $j$ to treat the next cohort of |
| 57 | patients unless the RDS of dose level $j$ is "E," at which point terminate the |
| 58 | trial. In the event of Case A or Case B, to prevent getting stuck in a local |
| 59 | dose, an extra dose exploration rule is implemented to escalate to the next |
| 60 | higher untried dose if the following two conditions are met: |
| 61 | ○ The number of patients treated at the current dose is $\ge 15$ . |
| 62 | o The next higher dose is not eliminated and has never been used for |
| 63 | treating patients. |

3. Repeat step 2 until the maximum sample size of 60 is reached or if the number of patients treated on any dose reaches 20. Then, use the isotonic estimation method described in Lin et al. 1 to select the OBD as the dose that is admissible and that has the highest estimated utility.



**Figure 1.** Flowchart for trial conduct using the BOIN12 design, where N\*=5, and  $(\lambda e, \lambda d) = (0.118, 0.179)$ .

**eTable 1.** Rank-based desirability score (RDS) table for the BOIN12 design, where "E" means elimination. A larger value of RDS means higher desirability, and any value of RDS is deemed higher than "E". **#Pts** denotes the number of evaluable patients treated at current dose; **#Tox** denotes the number of evaluable patients who experience efficacy.

| #Pts | #Tox | #Ef | f RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 0 | 0 | 0 | 262 | 15 | 0 | 7 | 96 | 15 | 4 | 9 | 61 | 20 | 2 | 19 | 528 |
| 5 | 0 | <= 1 | Е | 15 | 0 | 8 | 159 | 15 | 4 | 10 | 115 | 20 | 2 | 20 | 556 |
| 5 | 0 | 2 | 169 | 15 | 0 | 9 | 232 | 15 | 4 | 11 | 183 | 20 | 3 | <= 9 | E |
| 5 | 0 | 3 | 268 | 15 | 0 | 10 | 297 | 15 | 4 | 12 | 256 | 20 | 3 | 10 | 19 |
| 5 | 0 | 4 | 377 | 15 | 0 | 11 | 366 | 15 | 4 | 13 | 321 | 20 | 3 | 11 | 47 |
| 5 | 0 | 5 | 483 | 15 | 0 | 12 | 435 | 15 | 4 | 14 | 389 | 20 | 3 | 12 | 90 |

| #Pts | #Tox | #Ef | f RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 5 | 1 | <= 1 | E | 15 | 0 | 13 | 497 | 15 | 4 | 15 | 457 | 20 | 3 | 13 | 147 |
| 5 | 1 | 2 | 101 | 15 | 0 | 14 | 542 | 15 | >= 5 | Any | Е | 20 | 3 | 14 | 213 |
| 5 | 1 | 3 | 199 | 15 | 0 | 15 | 565 | 20 | 0 | <= 9 | E | 20 | 3 | 15 | 264 |
| 5 | 1 | 4 | 308 | 15 | 1 | <= 6 | E | 20 | 0 | 10 | 90 | 20 | 3 | 16 | 328 |
| 5 | 1 | 5 | 413 | 15 | 1 | 7 | 61 | 20 | 0 | 11 | 147 | 20 | 3 | 17 | 391 |
| 5 | >= 2 | Any | E | 15 | 1 | 8 | 115 | 20 | 0 | 12 | 213 | 20 | 3 | 18 | 448 |
| 10 | 0 | <= 4 | Е | 15 | 1 | 9 | 183 | 20 | 0 | 13 | 264 | 20 | 3 | 19 | 501 |
| 10 | 0 | 5 | 172 | 15 | 1 | 10 | 256 | 20 | 0 | 14 | 328 | 20 | 3 | 20 | 539 |

| #Pts | #Tox | #E | ff RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 10 | 0 | 6 | 250 | 15 | 1 | 11 | 321 | 20 | 0 | 15 | 391 | 20 | 4 | <= 9 | E |
| 10 | 0 | 7 | 330 | 15 | 1 | 12 | 389 | 20 | 0 | 16 | 448 | 20 | 4 | 10 | 8 |
| 10 | 0 | 8 | 414 | 15 | 1 | 13 | 457 | 20 | 0 | 17 | 501 | 20 | 4 | 11 | 27 |
| 10 | 0 | 9 | 492 | 15 | 1 | 14 | 514 | 20 | 0 | 18 | 539 | 20 | 4 | 12 | 59 |
| 10 | 0 | 10 | 545 | 15 | 1 | 15 | 550 | 20 | 0 | 19 | 561 | 20 | 4 | 13 | 109 |
| 10 | 1 | <= 4 | Е | 15 | 2 | <= 6 | E | 20 | 0 | 20 | 571 | 20 | 4 | 14 | 170 |
| 10 | 1 | 5 | 117 | 15 | 2 | 7 | 31 | 20 | 1 | <= 9 | E | 20 | 4 | 15 | 227 |
| 10 | 1 | 6 | 196 | 15 | 2 | 8 | 75 | 20 | 1 | 10 | 59 | 20 | 4 | 16 | 287 |

| #Pts | #Tox | #Et | ff RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 10 | 1 | 7 | 286 | 15 | 2 | 9 | 136 | 20 | 1 | 11 | 109 | 20 | 4 | 17 | 351 |
| 10 | 1 | 8 | 360 | 15 | 2 | 10 | 204 | 20 | 1 | 12 | 170 | 20 | 4 | 18 | 410 |
| 10 | 1 | 9 | 444 | 15 | 2 | 11 | 276 | 20 | 1 | 13 | 227 | 20 | 4 | 19 | 468 |
| 10 | 1 | 10 | 513 | 15 | 2 | 12 | 347 | 20 | 1 | 14 | 287 | 20 | 4 | 20 | 515 |
| 10 | 2 | <= 4 | Е | 15 | 2 | 13 | 412 | 20 | 1 | 15 | 351 | 20 | 5 | <= 9 | E |
| 10 | 2 | 5 | 69 | 15 | 2 | 14 | 478 | 20 | 1 | 16 | 410 | 20 | 5 | 10 | 2 |
| 10 | 2 | 6 | 141 | 15 | 2 | 15 | 529 | 20 | 1 | 17 | 468 | 20 | 5 | 11 | 12 |
| 10 | 2 | 7 | 220 | 15 | 3 | <= 6 | E | 20 | 1 | 18 | 515 | 20 | 5 | 12 | 34 |

| #Pts | #Tox | #E1 | ff RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 10 | 2 | 8 | 306 | 15 | 3 | 7 | 16 | 20 | 1 | 19 | 549 | 20 | 5 | 13 | 73 |
| 10 | 2 | 9 | 387 | 15 | 3 | 8 | 46 | 20 | 1 | 20 | 566 | 20 | 5 | 14 | 129 |
| 10 | 2 | 10 | 467 | 15 | 3 | 9 | 96 | 20 | 2 | <= 9 | Е | 20 | 5 | 15 | 192 |
| 10 | 3 | <= 4 | Е | 15 | 3 | 10 | 159 | 20 | 2 | 10 | 34 | 20 | 5 | 16 | 243 |
| 10 | 3 | 5 | 37 | 15 | 3 | 11 | 232 | 20 | 2 | 11 | 73 | 20 | 5 | 17 | 312 |
| 10 | 3 | 6 | 94 | 15 | 3 | 12 | 297 | 20 | 2 | 12 | 129 | 20 | 5 | 18 | 371 |
| 10 | 3 | 7 | 172 | 15 | 3 | 13 | 366 | 20 | 2 | 13 | 192 | 20 | 5 | 19 | 430 |
| 10 | 3 | 8 | 250 | 15 | 3 | 14 | 435 | 20 | 2 | 14 | 243 | 20 | 5 | 20 | 488 |

| #Pts | #Tox | #Ef | f RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS | #Pts | #Tox | #Eff | RDS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | , | | | | | | | |
| 10 | 3 | 9 | 330 | 15 | 3 | 15 | 497 | 20 | 2 | 15 | 312 | 20 | >=<br>6 | Any | E |
| 10 | 3 | 10 | 414 | 15 | 4 | <= 6 | E | 20 | 2 | 16 | 371 | | | | |
| 10 | >= 4 | Any | E | 15 | 4 | 7 | 6 | 20 | 2 | 17 | 430 | | | | |
| 15 | 0 | <= 6 | E | 15 | 4 | 8 | 23 | 20 | 2 | 18 | 488 | | | | |

#### Reference

- 1. Lin R., Zhou Y., Yan, F., Li D., and Yuan, Y. (2020). BOIN12: Bayesian optimal interval Phase I/II trial design for utility-based dose finding with immunotherapy and targeted therapies, *JCO Precision Oncology 4*, 1393-1402.
- 2. Zhou, Y., Lin, R., Kuo, Y., Lee, J. J, & Yuan, Y. (2021). BOIN suite: a software platform to design and implement novel early phase clinical trials. *JCO Clinical Cancer Informatics* 5, 91-101.